CLINICAL TRIAL: NCT06798519
Title: A Relative Bioavailability Study of HNC364 Following Intramuscular Injections Vs. AZILECT® (Rasagiline Tablet) Following Oral Administration At the Steady-State in Healthy Adult Subjects
Brief Title: Relative Bioavailability Study of HNC364 Injectable Suspension
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Henovcom Bioscience Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNC364-A102
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease (PD)
MeSH Terms: interventions — rasagiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HNC364 Injectable Suspension (Experimental): Subjects in HNC364 cohort will receive a deep IM injection of HNC364 injectable suspension in the deltoid muscle at a dose of 60 mg every 4 weeks for 4 repeated doses. Subjects will be allowed to leave the clinical site the next day after receiving each dose and return to clinical site on 7 days, 14 days and 28 days (before next administration) after each dose for safety and tolerability assessments. Besides, subjects will return to the clinical site on 4 days after the first dose and the last dose due to PK and PD blood sample collections.
  Interventions: Drug: HNC364 Injectable Suspension
- Rasagiline Tablets (Active Comparator): Subjects in rasagiline tablets cohort will receive 1 mg of rasagiline tablets orally once daily for 20 days, followed by 2 mg once daily for 5 days. Subjects will remain domiciled at the clinic stay until Day 26 and have a follow-up visit on Day 29 due to PK and PD blood sample collections
  Interventions: Drug: Rasagiline Tablets

INTERVENTIONS:
Drug: HNC364 Injectable Suspension — Subjects in HNC364 cohort will receive a deep IM injection of HNC364 injectable suspension in the deltoid muscle at a dose of 60 mg every 4 weeks for 4 repeated doses. Subjects will be allowed to leave the clinical site the next day after receiving each dose and return to clinical site on 7 days, 14 days and 28 days (before next administration) after each dose for safety and tolerability assessments. Besides, subjects will return to the clinical site on 4 days after the first dose and the last dose due to PK and PD blood sample collections.
  Arms: HNC364 Injectable Suspension
Drug: Rasagiline Tablets — Subjects in rasagiline tablets cohort will receive 1 mg of rasagiline tablets orally once daily for 20 days, followed by 2 mg once daily for 5 days. Subjects will remain domiciled at the clinic stay until Day 26 and have a follow-up visit on Day 29 due to PK and PD blood sample collections
  Arms: Rasagiline Tablets

SUMMARY:
HNC364 is a new pro-drug of rasagiline as a long-acting injection for deep IM deltoid injection, for the treatment of Parkinson"s disease (PD). As a pro-drug of rasagiline, HNC364 will readily and completely convert to rasagiline after the IM administration.

This is a non-randomized, open-label, Phase 1 study to evaluate the relative bioavailability of HNC364 injectable suspension relative to AZILECT® (rasagiline tablets), to assess the safety and tolerability of multiple IM dose HNC364 injectable suspension dose administration in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements, and restrictions of the study. Are capable of giving informed consent and complying with study procedures.
2. Refer to Section 6.4 (all sub-sections) for full details regarding study restrictions and requirements.
3. Be able to complete the study according to the requirements of the study protocol.
4. Healthy adult subjects aged 18-55 (including boundary value), both male and female.
5. The body weight of male subjects shall not be less than 50 kg and that of female subjects shall not be less than 45 kg. BMI = body weight (kg)/height2 (M2), and the body mass index is in the range of 18 ~ 32 kg/m2 (including the critical value).
6. Vital signs, physical examination, laboratory tests, and electrocardiogram, etc. are normal, or abnormal results are judged by the Investigator to be clinically insignificant.
7. Nonsmoker, those who did not use other nicotine-containing products, those who quit smoking or stopped using other nicotine-containing products 3 months before the study drug administration.
8. Female or male subjects with potential fertility must agree to use an effective contraceptive method from the start of signing informed consent form until 6 months after the study drug administration to avoid pregnancy or make their partner pregnant.

Exclusion Criteria:

1. Prior to screening, subjects had clinically significant disease history as determined by the Investigator, including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immunological, psychiatric, cardio cerebrovascular disease or any reported history of sleep disorder.
2. Any history of suicide or at high risk for suicide assessment at screening.
3. The subject has a history of severe allergy or allergy to the study drug and any of its components or related excipients.
4. Prior to screening, those who have a history of gastrointestinal, liver and kidney diseases or surgery that potentially affect the absorption, distribution, metabolism and excretion of the study drug (except for uncomplicated appendectomy and hernia repair).
5. A history of alcoholism (alcoholism is defined as drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, 25 mL of spirits, or 100 mL of wine) or positive alcohol breath test during the screening period.
6. Those who had a history of drug abuse or used drugs within 2 years before screening or those who were positive for urinary drug screening during the screening period.
7. Subjects who had a history of smoking or used other nicotine-containing products within 3 months before the study drug administration, or who were positive for urine nicotine test during screening.
8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
9. Strong inhibitors and/or inducers of liver metabolizing enzymes (CYP1A2, 2A6, 2C8, 2C19, 3A4 and 3A5), strong inhibitors of liver metabolizing enzymes such as ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, acerbicin, etc., and strong inducers of liver metabolizing enzymes such as rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc. were used within 4 weeks before the study drug administration.
10. Any prescription drug, over-the-counter drug, any vitamin product or Chinese herbal medicine used within 2 weeks before the study drug administration.
11. Had consumed a special diet (including pitaya, mango, grapefruit, or certain foods containing high amounts of tyramine, etc.) or had vigorous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc., within 2 weeks before the administration.
12. Had consumed chocolate, any food or beverage containing caffeine or xanthine-rich within 72 hours before the study drug administration.
13. Taking any alcoholic product within 48 hours before the administration.
14. Donation of plasma within 30 days, or donation of blood or massive blood loss (≥ 400 mL) within 60 days, or donation of bone marrow or peripheral stem cells within 90 days before the study drug administration.
15. Participated in other clinical trials within 30 days prior to study drug administration.
16. Acute disease or concomitant medication from the signing of informed consent form to the study drug administration.
17. Lactating women or those with positive serum pregnancy results.
18. The researchers believe that subjects with other factors that are not suitable to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from time 0 to dose interval (AUCτ) | Day 1 to 56 days post dose
  The relative bioavailability of HNC364 injectable suspension and rasagiline tablets at the steady-state will be calculated by comparing the following PK parameters of rasagiline in both formulations.
  Due to the negligible plasma concentrations of HNC364 observed following intramuscular injection, the relative bioavailability calculations will be based on the assumption of complete conversion of HNC364 to rasagiline in vivo. To facilitate this comparison, the administered dose of HNC364 (60 mg) will be converted to an equivalent dose of rasagiline based on their respective molecular weights: 60 mg * 171.24 / 624.91 = 16.44 mg.
Number of Participants With Treatment Emergent Adverse Events | Day 1 to 56 days post dose
  The following assessments will be used to evaluate the safety of HNC364 and rasagiline: monitoring and assessment of adverse events (AEs) and concomitant medications; 12-lead electrocardiograms (ECGs); vital sign measurements (including blood pressure, heart rate, respiratory rate, and oral temperature); clinical laboratory test results (including serum chemistry, hematology, coagulation, and urinalysis); physical examinations and injection site reactions.

SECONDARY OUTCOMES:
maximum observed concentration (Cmax) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14.
  Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56.
  rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2.
  Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21.
  Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
time to maximum concentration (Tmax) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Time at which half the drug has been eliminated (t½) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Mean residence time (MRT) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Apparent total clearance for extravascular administration (CL/F) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Apparent volume of distribution during terminal phase (Vz/F) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Elimination rate constant (Kel) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Steady-state trough concentration (Css_min) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Average steady-state blood drug concentration (Css-av) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Steady-state peak concentration (Css_min) | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)
Platelet MAO-B activity | Day 1 to 56 days post dose
  HNC364 cohorts Dose 1: Pre dose (within 60 min); post dose at 4 (±5 min) and 24 (±60 min) hour; post dose at Days 4, 7, 10 and 14. Dose 2 and 3: Pre dose (within 60 min) Dose 4: Pre dose (within 60 min); post dose at 24 hour (±60 min); post dose at Days 4, 7, 10, 14, 29 and 56. rasagiline tablets cohort Study Day 1: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 1 should be taken before dosing on Days 2. Study Day 4: pre dose (up to 30 min); Study Day 7: pre dose (up to 30 min) and 1 hours (±1 min) post dose Study Days 10 and 14: pre dose (up to 30 min); Study Day 20: pre dose (up to 30 min) and 0.5, 1 hour (±1 min), 2, 4 hours (±2 min), 6, 12 hours (±5 min) and 24 hours (±30 min) post dose. The 24 hour post dose blood PK samples for Days 20 should be taken before dosing on Days 21. Study Day 21: 1 hours (±1 min) post dose Study Day 25: pre dose (up to 30 min)

IPD SHARING:
Plan to Share IPD: No